CLINICAL TRIAL: NCT07240376
Title: Efficacy and Safety of Stapokibart (CM310) in Non-Allergic Rhinitis With Eosinophilia Syndrome (ESSNARES): An Investigator-initiated, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of Stapokibart in Non-Allergic Rhinitis With Eosinophilia Syndrome
Acronym: ESSNARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Zheng Liu, M.D., Ph.D., FAAAAI Vice President, Chinese Society of Allergy Professor of Otolaryngology-Head & Neck Surgery Party Secretary of Zhongnan Hospital Wuhan University, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-NARES
Record Dates: First submitted 2025-09-30; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Non-Allergic Rhinitis With Eosinophilia Syndrome
Keywords: Stapokibart; Non-Allergic Rhinitis with Eosinophilia Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 group (Experimental): After enrollment, paticipants were given CM310 (with an initial dose of 600 mg followed by 300mg subcutaneous injection, once every two weeks) for 12 weeks. Follow up for another 8 weeks.Mometasone furoate was nasal sprayed daily during treatment
  Interventions: Biological: Stapokibart (CM310)
- Placebo group (Placebo Comparator): After enrollment, paticipants were given a placebo (subcutaneous injection, with the same dose as the experimental group, once every two weeks) for 12 weeks. Follow up for another 8 weeks. During the treatment period, mometasone furoate was sprayed nasal every day
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Stapokibart (CM310) — Paticipants were given CM310 (with an initial dose of 600 mg followed by 300mg subcutaneous injection, once every two weeks) for 12 weeks. Follow up for another 8 weeks.During the treatment period, mometasone furoate was sprayed nasal every day
  Arms: CM310 group
Other: Placebo — After enrollment, paticipants were given a placebo (subcutaneous injection, with the same dose as the experimental group, once every two weeks) for 12 weeks. Follow up for another 8 weeks. During the treatment period, mometasone furoate was sprayed nasal every day
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to learn if Stapokibart (CM310) works to treat Non-Allergic Rhinitis with Eosinophilia Syndrome (NARES) in adults. It will also learn about the safety of CM310.

The main questions it aims to answer are:

Does drug CM310 relieve the symptoms of participants? What medical problems do participants have when injecting CM310? Researchers will compare CM310 to a placebo (a look-alike substance that contains no drug) to see if CM310 works to treat NARES.

Participants will:

Inject CM310 or a placebo every 2 weeks for 12 weeks, and follow up for another 8 weeks.

Visit the clinic once every 2 weeks for checkups and tests. Keep a diary of their symptoms every day.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the efficacy of Stapokibart (CM310) in alleviating nasal and ocular symptoms, as well as its safety profile, in adult patients with Non-Allergic Rhinitis with Eosinophilia Syndrome (NARES) who have shown a suboptimal response to intranasal corticosteroids.

Adult NARES patients with an inadequate response to mometasone furoate nasal spray will be enrolled. While continuing treatment with intranasal mometasone furoate, patients will be randomized to receive either Stapokibart or a placebo. Over the 12-week treatment period and the subsequent 8-week follow-up period, the alleviation of nasal and ocular symptoms, the incidence of adverse events, and the results of safety assessments (such as physical examinations, electrocardiograms, complete blood counts, and blood biochemistry) will be evaluated. The final aim is to assess the efficacy and safety of Stapokibart in treating patients with NARES.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for participation in this clinical trial.

  1. The subject must understand the investigational nature of this study and must provide written informed consent, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to undergoing any study-related procedures.
  2. Aged ≥18 and ≤65 years, regardless of gender.
  3. Diagnosed with Non-Allergic Rhinitis with Eosinophilia Syndrome (NARES) according to the following criteria: chronic course lasting ≥2 years, with intermittent nasal symptoms including alternating nasal congestion, watery rhinorrhea, paroxysmal sneezing, nasal itching, postnasal drip, and hyposmia; with evidence against allergic rhinitis.
  4. Laboratory evidence: negative serum Specific Immunoglobulin E (sIgE) and negative Skin Prick Test (SPT); nasal secretion eosinophil proportion >20% (after excluding epithelial cells).
  5. The subject's history prior to the screening period indicates inadequate control of NARES symptoms (with an iTNSS ≥4 and at least one of the symptoms - nasal congestion, rhinorrhea, nasal itching, or sneezing - scoring ≥2) despite the use of intranasal corticosteroids or other medications (e.g., antihistamines, leukotriene receptor antagonists) following symptom onset.
  6. At the baseline visit (after run-in treatment), the subject must meet the following criteria: an iTNSS ≥4, the average of the most recent 6 daily Reflective Total Nasal Symptom Scores (rTNSS) ≥4, and at least one of the symptoms - nasal congestion, rhinorrhea, nasal itching, or sneezing - scoring ≥2 in these assessments (i.e., the 3 morning and 3 evening evaluations over the last three 24-hour periods, including the iTNSS assessment at the baseline visit).
  7. Willing and able to comply with all visits, study-related procedures, and questionnaires, including adherence to required background medications and completion of a daily electronic diary (eDiary). During the screening/run-in period, subjects must complete at least 80% of the diary assessments.
  8. Subjects agree to use highly effective contraception (including vasectomy, abstinence, etc.) throughout the study period (from signing the ICF until 3 months after the last dose of study drug).

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible to participate in this clinical trial.

  1. History of allergy to study drugs: hypersensitivity or intolerance to mometasone furoate, loratadine, CM310 injection, or any component of the placebo.
  2. Laboratory abnormalities: severe hepatic or renal dysfunction, abnormal liver function [Alanine Aminotransferase (ALT)/Aspartate Transaminase (AST) >1.5 × Upper Limit of Normal (ULN), or Total Bilirubin (TBIL) >1.5 × ULN with abnormal AST] or abnormal renal function (serum creatinine >1.2 × ULN); clinically significant abnormalities in laboratory blood chemistry or hematology results at screening (Visit 1) or baseline (Visit 2) as judged by the investigator.
  3. History of harmful behavior: history of drug abuse, alcohol dependence (average daily alcohol intake >40 g) within 2 years prior to screening, or current drug user.
  4. Currently receiving allergen immunotherapy (subcutaneous or sublingual immunotherapy [SCIT/SLIT]). Subjects who discontinued SCIT/SLIT ≥3 years prior to randomization and are not on a maintenance regimen are eligible.
  5. Use of any rescue medication during the screening and run-in periods.
  6. Nasal procedure history at screening (Visit 1): nasal sinus surgery within 1 year prior to screening or presence of unhealed nasal trauma.
  7. Drug exposure at screening (Visit 1): participation in another drug clinical trial and use of an investigational drug within 3 months prior to screening, or planned use of another investigational drug during the study.
  8. Vaccination at screening (Visit 1): receipt of a live attenuated vaccine within 12 weeks prior to screening or planned vaccination with a live attenuated vaccine during the trial.
  9. Ocular disease at screening (Visit 1): presence of glaucoma, cataract, ocular herpes simplex, infectious conjunctivitis, or other ocular infections.
  10. Infection history at screening (Visit 1): active or inactive pulmonary tuberculosis infection; untreated localized or systemic fungal, bacterial, viral, or parasitic infection requiring ongoing treatment which, in the investigator's judgment, may place the subject at undue risk or affect result interpretation (e.g., severe infection requiring hospitalization and/or IV or equivalent oral antibiotics); symptomatic herpes zoster infection not resolved at screening; recurrent infections (including but not limited to recurrent cellulitis, chronic osteomyelitis). Subjects with only recurrent, mild, uncomplicated herpes labialis and/or genital herpes may be enrolled. Subjects with a history of active or latent tuberculosis with written evidence of adequate treatment, no history of re-exposure since completion of treatment, and no evidence of active tuberculosis on chest X-ray at screening may be enrolled.
  11. Subjects with comorbid asthma (including suspected asthma) are excluded if they meet any of the following: FEV1 ≤60% of predicted; or an asthma exacerbation within 3 months prior to screening requiring systemic corticosteroids or hospitalization (>24 hours); or required inhaled corticosteroid dosage >1000 μg fluticasone propionate or equivalent.
  12. Known history of recurrent acute or chronic rhinosinusitis, defined as requiring systemic antibiotic treatment within 3 months prior to screening, or >4 recurrences within 2 years prior to screening.
  13. Conditions affecting drug deposition: nasal disease or symptoms/signs identified during screening or prior to randomization that, in the investigator's judgment, may affect intranasal drug deposition, such as acute or chronic sinusitis, symptoms/signs of chronic purulent postnasal drip, rhinitis medicamentosa, nasal polyps, vasomotor rhinitis, other clinically significant respiratory tract deformities/nasal structural abnormalities, significant nasal trauma (e.g., penetrating injury), or significant nasal septum deviation; any nasal mucosal erosion, nasal septum ulcer, or perforation at screening or prior to randomization; recent nasal piercing not fully healed that may cause nasal symptoms, or planned new nasal piercing during the study.
  14. Restricted medication use prior to run-in period: use of the following medications and/or treatments within a specified time prior to the run-in period or within 5 half-lives of the drug: IL-4Rα antagonists (within 10 weeks or 5 half-lives), vasoconstrictors (3 days), strong sedatives (3 days), antihistamines (10 days), decongestants (3 days), leukotriene receptor antagonists (7 days), anticholinergics (7 days), cromolyn-like drugs (14 days), systemic antibiotics (14 days), ocular mast cell stabilizers (14 days), monoamine oxidase inhibitors (14 days), tricyclic antidepressants (14 days), strong CYP3A4 inducers/inhibitors (14 days), anti-allergy Chinese herbal medicines (14 days), short- or medium-acting systemic corticosteroids (4 weeks), long-acting systemic corticosteroids (6 weeks), immunotherapy such as desensitization therapy and other biologic monoclonal antibody therapies (3 months), etc.
  15. Immunosuppression: treatment with biologics/systemic immunosuppressants (including but not limited to methotrexate, cyclosporine, mycophenolate mofetil, tacrolimus, penicillamine, sulfasalazine, hydroxychloroquine, azathioprine, cyclophosphamide) for inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cholangitis, systemic lupus erythematosus, multiple sclerosis) within 8 weeks prior to randomization or within 5 half-lives (whichever is longer); known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) even if resolved; or abnormally frequent, recurrent, or prolonged infections as judged by the investigator.
  16. Restricted medication use during the trial: planned use during the trial of the following drugs and/or treatments: a. strong CYP3A4 inducers/inhibitors; b. chronic or intermittent use of corticosteroids (except investigational product); c. antihistamines; d. leukotriene receptor antagonists; e. mast cell membrane stabilizers; f. systemic or intranasal decongestants; g. anticholinergics; h. immunosuppressants; i. anti-allergy Chinese herbal medicines/proprietary Chinese medicines/health products; j. anti-IgE antibodies (e.g., omalizumab for injection); k. nasal irrigations (including saline).
  17. Female subjects who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.
  18. Presence of any other medical or psychological condition that, in the investigator's opinion, may indicate a new and/or insufficiently understood disease, participation in this clinical study may pose an unreasonable risk to the subject, may make the subject unable to participate stably in the study, or may interfere with study evaluations.
  19. Geographical restrictions: planned long-term travel away from the place of residence for ≥4 consecutive weeks during the trial, or planned residence in an area with a significantly different climate from the long-term place of residence.
  20. Previous participation in a CM310 clinical trial.
  21. Previous use of any anti-IL-4Rα monoclonal antibody (e.g., dupilumab) with inadequate treatment response (e.g., treatment failure or intolerance).
  22. Presence of other uncontrolled severe diseases or recurrent chronic comorbidities, including but not limited to active infection, cardiovascular and cerebrovascular diseases, tuberculosis or other pathogen infections, diabetes, autoimmune diseases, human immunodeficiency virus (HIV) infection, Treponema pallidum infection, active hepatitis B or C, or parasitic diseases.
  23. History of malignancy within 5 years prior to screening.
  24. Any other medical or non-medical condition that, in the investigator's opinion, makes the subject unsuitable for participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline in the Reflective Total Nasal Symptom Score (rTNSS) at Week 12. | From enrollment to the end of treatment at 12 weeks
  The Reflective Total Nasal Symptom Score （rTNSS） assesses the severity of nasal symptoms over the past 12 hours and is evaluated in the morning (ante meridiem rTNSS, AMrTNSS) and evening (post meridiem rTNSS, PMrTNSS). The daily rTNSS is the average of AMrTNSS and PMrTNSS. rTNSS isa scoring scale ranging from 0 to 12, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
reflective Total Nasal Symptom Scores | From enrollment to the end of study at 20 weeks
  Mean change from baseline in daily morning AM reflective Total Nasal Symptom Scores (AMrTNSS) during the treatment period; Mean change from baseline in daily evening PM reflective Total Nasal Symptom Scores (PMrTNSS) during the treatment period; rTNSS is the mean of AMrTNSS and PMrTNSS. The rTNSS, AMrTNSS, PMrTNSS are scoring scales ranging from 0 to 12, with higher scores indicating more severe symptoms
Instant Total Nasal Symptom Score (iTNSS) | From enrollment to the end of study at 20 weeks
  Mean change from baseline in the Instant Total Nasal Symptom Score (iTNSS) immediately prior to dosing during the treatment period; The iTNSS is a scoring scale ranging from 0 to 12, with higher scores indicating more severe symptoms
reflective individual nasal symptom scores | From enrollment to the end of study at 20 weeks
  Mean change from baseline in daily reflective individual nasal symptom scores (rhinorrhea, nasal congestion, nasal itching, sneezing) during the treatment period. Daily reflective individual nasal symptom scores are the means of daily daytime (AM) reflective individual nasal symptom scores and daily nighttime (PM) reflective individual nasal symptom scores.
  Each symptom score is a scale ranging from 0 to 3, with higher scores indicating more severe symptoms
Reflective Total Ocular Symptom Score | From enrollment to the end of study at 20 weeks
  Mean change from baseline in the daily morning ante meridiem rTOSS (AMrTOSS) during the treatment period should be recorded; and mean change from baseline in the daily evening post meridiem rTOSS (PMrTOSS) during the treatment period should be recored; Mean change from baseline in the daily Reflective Total Ocular Symptom Score (rTOSS) during the treatment period should be calculated. Daily rTOSS is the mean of AMrTOSS and daily PMrTOSS.
  The rTOSS, AMrTOSS, PMrTOSS are scoring scales ranging from 0 to 9, with higher scores indicating more severe symptoms
Instant Total Ocular Symptom Score (iTOSS) | From enrollment to the end of study at 20 weeks
  Mean change from baseline in the Instant Total Ocular Symptom Score (iTOSS) immediately prior to dosing during the treatment period.
  The rTOSS is a scoring scale ranging from 0 to 9, with higher scores indicating more severe symptoms
reflective individual ocular symptom scores | From enrollment to the end of study at 20 weeks
  Mean change from baseline in daily reflective individual ocular symptom scores (ocular itching, tearing, eye redness) during the treatment period.
  Daily reflective individual ocular symptom scores are means of daytime (AM) reflective individual ocular symptom scores and nighttime (PM) reflective individual ocular symptom scores.
  Each of reflective individual ocular symptom score is a scale ranging from 0 to 3, with higher scores indicating more severe symptoms.
Assessment of patient quality of life using the Rhino-Conjunctivitis Quality of Life Questionnaire (RQLQ) | From enrollment to the end of study at 20 weeks
  Assessment of patient quality of life using the Rhino-Conjunctivitis Quality of Life Questionnaire (RQLQ), including domains such as daily activities, sleep disturbance, practical problems, nasal symptoms, ocular symptoms, and emotional function, with calculation of the total score.
  The RQLQ is a scoring scale ranging from 0 to 168, with higher scores indicating a greater impact of symptoms on daily life.
visual analogue scale of olfactory function | From enrollment to the end of treatment at 12 weeks
  Evaluation of olfactory function using the visual analogue scale (VAS).The VAS is a scoring scale ranging from 0 to 10, with higher scores indicating more severe symptoms.
Overall evaluation of treatment response | From enrollment to the end of the study at 20 weeks
  Overall evaluation of treatment response based on a 7-point categorical scale, where subjects rate the change in NARES symptoms at the end of the study as follows: significantly improved, moderately improved, mildly improved, no change, mildly worsened, moderately worsened, or significantly worsened.

OTHER OUTCOMES:
Area Under the Curve (AUC) for the change from baseline in daily rTNSS during the treatment period. | From enrollment to the end of treatment at 12 weeks
  Area Under the Curve (AUC) for the change from baseline in daily rTNSS during the treatment period.
Number of days with no or mild symptoms during the treatment period. | From enrollment to the end of treatment at 12 weeks
  For daily rTNSS and rTOSS, days with no or mild symptoms are defined as follows:
  No or mild nasal symptoms: each individual symptom score (rhinorrhea, nasal congestion, nasal itching, sneezing) ≤ 1.
  No or mild ocular symptoms: each individual symptom score (ocular itching, tearing, eye redness) ≤ 1.
Peripheral Blood eosinophil | At day 1, day 85 and day 141
  Peripheral Blood Parameters: Changes in eosinophil count will be recorded and Changes in eosinophil percentage will be calculated
Peripheral Blood Cytokines and chemokines | At day 1, day 85 and day 141
  Peripheral Blood Cytokines and chemokines will be detected: Interleukin (IL)-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17A, Tumor Necrosis Factor (TNF)-α, Interferon (IFN)-γ, Monocyte Chemoattractant Protein (MCP)-1, Granulocyte Colony-Stimulating Factor (G-CSF), Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), Eosinophil Cationic Protein (ECP).
  The levels of peripheral blood cytokines and chemokines will be represented in picogram/milligram or nanogram/milligram
Peripheral Blood Immunoglobulins | At day 1, day 85 and day 141
  Concentrations of specific and total Immunoglobulin (Ig) A, IgG4, IgG, IgE, and total IgM will be detected and represented in picogram/milligram or nanogram/milligram
Nasal Secretion Neurotransmitters and Proteases | At day 1, day 85 and day 141
  Nasal secretion neurotransmitters and proteases: Vasoactive Intestinal Polypeptide (VIP), Substance P, histamine, 5-Hydroxytryptamine (5-HT), tryptase will be detected.The levels of neurotransmitters and proteases will be represented in picogram/milligram or nanogram/milligram
Nasal Secretion Cytokines and chemokines | At day 1, day 85 and day 141
  Nasal Secretion cytokines and chemokines:IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17A, TNF-α, IFN-γ, MCP-1, G-CSF, GM-CSF, ECP, Charcot-Leyden Crystal (CLC), eotaxin-1, eotaxin-2 will be detected.
  The levels of nasal secretion cytokines and chemokines will be represented in picogram/milligram or nanogram/milligram
Nasal Brush Cytology | At day 1, day 85 and day 141
  Nasal brush cytology: changes in eosinophil count will be recorded and changes in eosinophil percentage will be calculated.
mRNA expression levels of genes of nasal brush cells | At day 1, day 85 and day 141
  The mRNA expression levels of CLC, Arachidonate 15-Lipoxygenase (ALOX15), ALOX5, Cyclooxygenase (COX), Transient Receptor Potential Melastatin 8 (TRPM8), Transient Receptor Potential Vanilloid subfamily 1 (TRPV1), TRPV4, and Transient Receptor Potential Ankyrin subtype 1 protein (TRPA1) will be detected.
Safety Endpoints | From enrollment to the end of study at 20 weeks
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) will be reported
Safty endpoint | From enrollment to the end of study at 20 weeks
  Abnormalities in physical examinations
Safty endpoint | From enrollment to the end of study at 20 weeks
  Abnormalities in 12-lead electrocardiogram (ECG) will be reported
Safty endpoint | From enrollment to the end of study at 20 weeks
  Abnormalities in complete blood count, blood chemistry, urinalysis will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Principal Investigator — Zhongnan Hospital
Locations (11):
- China (11):
  - Clifford Hospital, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji hospital, Tongji medical college, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Provincial Hospital of Integrated Chinese and Western Medicine, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Eye & Ent Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 3 years after the publication of results
Access Criteria: The study protocol, statistical analysis plan, and study results from this research will be available on ClinicalTrials.gov and in journals where the primary results are published. If additional data is required by other researchers, they may contact the corresponding author to request access to the data after the publication of the primary study findings.